CLINICAL TRIAL: NCT04554693
Title: The Use of Low Dose Metronidazole to Decrease Postoperative Pain After Endometriosis Surgery: a Prospective, Randomized, Placebo-Controlled Trial
Brief Title: The Use of Low Dose Metronidazole to Decrease Postoperative Pain After Endometriosis Surgery
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Resad Pasic, Director, Fellowship in Advanced Gynecologic Endoscopy, Department of Obstetrics and Gynecology and Woman's Health, University of Louisville School of Medicine, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200544
Record Dates: First submitted 2020-09-05; First posted 2020-09-18 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Endometriosis; Endometriosis-related Pain
MeSH Terms: conditions — Endometriosis | interventions — Metronidazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metronidazole (Experimental): Metronidazole
  Interventions: Drug: Metronidazole Oral
- Placebo (Placebo Comparator): Halal and Kosher certified gelatin placebo capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metronidazole Oral — 250 mg oral three times a day for 14 days
  Arms: Metronidazole
Drug: Placebo — Halal and Kosher certified gelatin placebo capsules oral three times a day for 14 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine a difference in participant reported pain after endometriosis surgery in participants given oral metronidazole versus placebo.

DETAILED DESCRIPTION:
The study is a prospective, randomized, placebo-controlled trial. Women scheduled for endometriosis surgery between 18-50 years of age will be invited to participate in the study.

Participants with surgically staged endometriosis will be randomized to the metronidazole plus routine postoperative care arm or the placebo plus routine postoperative care arm. Participants will take study or placebo drug for a total of 14 days.

Participants will complete surveys at baseline and postoperatively at 6 weeks, 6 months, 1 year, 2 years, 3 years, 4 years, and 5 years reporting intensity of endometriosis associated pain on a visual analog scale, pregnancy outcomes, quality of life, and sexual health.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent
* Women aged 18-50 years old
* Scheduled to undergo excision of endometriosis
* Able to read and write in English and or Spanish
* Pain score > 2 on a 10 point visual analogue scale at baseline
* Negative screening by CAGE questionnaire

Exclusion Criteria:

* Refusal to surgery
* Contraindication to surgery
* Known allergy to metronidazole
* Known allergy to any component in gelatin placebo capsules
* Scheduled hysterectomy
* Endometriosis excision surgery within the last 3 months
* Elevated serum creatinine
* Abnormal liver function test greater than 2 times the normal
* Current pregnancy
* Breastfeeding
* Use of Disulfiram within the last 2 weeks
* History of Cockayne syndrome
* Inability to abstain from alcohol during the use of study drug

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female participants
Enrollment: 90 (Estimated)
Dates: Start 2020-10-19 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Self-reported pain persistence | 6 weeks postoperatively.
  The outcome of binary, subject pain persistence, assessed as yes or no, will be compared between groups using the Fisher exact test.

SECONDARY OUTCOMES:
Quality of life scores | 1 year postoperatively.
  Endometriosis Health Profile-5 on scale of 1-100 with higher scores meaning worse outcome
Quality of life scores | 6 months postoperatively.
  Endometriosis Health Profile-5 on scale of 1-100 with higher scores meaning worse outcome
Quality of life scores | 6 weeks postoperatively.
  Endometriosis Health Profile-5 on scale of 1-100 with higher scores meaning worse outcome
Quality of life scores | 5 years postoperatively.
  Endometriosis Health Profile-5 on scale of 1-100 with higher scores meaning worse outcome
Sexual health | 6 weeks postoperatively.
  Female sexual function index on a scale of 0-36 with higher scores meaning higher sexual dysfunction
Sexual health | 6 months postoperatively.
  Female sexual function index on a scale of 0-36 with higher scores meaning higher sexual dysfunction
Sexual health | 1 year postoperatively.
  Female sexual function index on a scale of 0-36 with higher scores meaning higher sexual dysfunction
Sexual health | 5 year postoperatively.
  Female sexual function index on a scale of 0-36 with higher scores meaning higher sexual dysfunction
Self-reported pain persistence | 1 year postoperatively.
  The outcome of binary, subject pain persistence, assessed as yes or no, will be compared between groups using the Fisher exact test.
Self-reported pain persistence | 6 months postoperatively.
  The outcome of binary, subject pain persistence, assessed as yes or no, will be compared between groups using the Fisher exact test.

OTHER OUTCOMES:
Fertility | 6 months postoperatively
  Number of pregnancies and miscarriages postoperatively will be compared
Fertility | 1 year postoperatively
  Number of pregnancies and miscarriages postoperatively will be compared
Fertility | 5 years postoperatively
  Number of pregnancies and miscarriages postoperatively will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Resad Pasic, MD, PhD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville Hospital, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burney RO, Giudice LC. Pathogenesis and pathophysiology of endometriosis. Fertil Steril. 2012 Sep;98(3):511-9. doi: 10.1016/j.fertnstert.2012.06.029. Epub 2012 Jul 20. PMID 22819144
- [Background] Working group of ESGE, ESHRE and WES; Saridogan E, Becker CM, Feki A, Grimbizis GF, Hummelshoj L, Keckstein J, Nisolle M, Tanos V, Ulrich UA, Vermeulen N, De Wilde RL. Recommendations for the Surgical Treatment of Endometriosis. Part 1: Ovarian Endometrioma. Hum Reprod Open. 2017 Dec 19;2017(4):hox016. doi: 10.1093/hropen/hox016. eCollection 2017. PMID 31486802
- [Background] Practice bulletin no. 114: management of endometriosis. Obstet Gynecol. 2010 Jul;116(1):223-236. doi: 10.1097/AOG.0b013e3181e8b073. No abstract available. PMID 20567196
- [Background] Abbott J, Hawe J, Hunter D, Holmes M, Finn P, Garry R. Laparoscopic excision of endometriosis: a randomized, placebo-controlled trial. Fertil Steril. 2004 Oct;82(4):878-84. doi: 10.1016/j.fertnstert.2004.03.046. PMID 15482763
- [Background] Sutton CJ, Ewen SP, Whitelaw N, Haines P. Prospective, randomized, double-blind, controlled trial of laser laparoscopy in the treatment of pelvic pain associated with minimal, mild, and moderate endometriosis. Fertil Steril. 1994 Oct;62(4):696-700. doi: 10.1016/s0015-0282(16)56990-8. PMID 7926075
- [Background] Quaranta G, Sanguinetti M, Masucci L. Fecal Microbiota Transplantation: A Potential Tool for Treatment of Human Female Reproductive Tract Diseases. Front Immunol. 2019 Nov 26;10:2653. doi: 10.3389/fimmu.2019.02653. eCollection 2019. PMID 31827467
- [Background] Leonardi M, Hicks C, El-Assaad F, El-Omar E, Condous G. Endometriosis and the microbiome: a systematic review. BJOG. 2020 Jan;127(2):239-249. doi: 10.1111/1471-0528.15916. Epub 2019 Sep 19. PMID 31454452
- [Background] Chadchan SB, Cheng M, Parnell LA, Yin Y, Schriefer A, Mysorekar IU, Kommagani R. Antibiotic therapy with metronidazole reduces endometriosis disease progression in mice: a potential role for gut microbiota. Hum Reprod. 2019 Jun 4;34(6):1106-1116. doi: 10.1093/humrep/dez041. PMID 31037294
- [Background] Simoens S, Hummelshoj L, D'Hooghe T. Endometriosis: cost estimates and methodological perspective. Hum Reprod Update. 2007 Jul-Aug;13(4):395-404. doi: 10.1093/humupd/dmm010. PMID 17584822
- [Background] Nogueira F, Sharghi S, Kuchler K, Lion T. Pathogenetic Impact of Bacterial-Fungal Interactions. Microorganisms. 2019 Oct 16;7(10):459. doi: 10.3390/microorganisms7100459. PMID 31623187
- [Background] Mert I, Walther-Antonio M, Mariani A. Case for a role of the microbiome in gynecologic cancers: Clinician's perspective. J Obstet Gynaecol Res. 2018 Sep;44(9):1693-1704. doi: 10.1111/jog.13701. Epub 2018 Aug 2. PMID 30069974
- [Background] Moloney RD, Johnson AC, O'Mahony SM, Dinan TG, Greenwood-Van Meerveld B, Cryan JF. Stress and the Microbiota-Gut-Brain Axis in Visceral Pain: Relevance to Irritable Bowel Syndrome. CNS Neurosci Ther. 2016 Feb;22(2):102-17. doi: 10.1111/cns.12490. Epub 2015 Dec 10. PMID 26662472
- [Background] Guo R, Chen LH, Xing C, Liu T. Pain regulation by gut microbiota: molecular mechanisms and therapeutic potential. Br J Anaesth. 2019 Nov;123(5):637-654. doi: 10.1016/j.bja.2019.07.026. Epub 2019 Sep 21. PMID 31551115
- [Background] Glick LR, Sossenheimer PH, Ollech JE, Cohen RD, Hyman NH, Hurst RD, Rubin DT. Low-Dose Metronidazole is Associated With a Decreased Rate of Endoscopic Recurrence of Crohn's Disease After Ileal Resection: A Retrospective Cohort Study. J Crohns Colitis. 2019 Sep 19;13(9):1158-1162. doi: 10.1093/ecco-jcc/jjz047. PMID 30809655